CLINICAL TRIAL: NCT06994780
Title: Lung Ultrasound Evaluation of the Effects of Positive End-Expiratory Pressure (PEEP) and Recruitment Strategies Adjusted for Intraoperative Dynamic Compliance on Postoperative Respiratory Complications in Obese Patients Planned for Laparoscopic Surgery
Brief Title: Lung Ultrasound Evaluation of the Effects of PEEP and Recruitment Strategies Adjusted for Intraoperative Dynamic Compliance on Postoperative Respiratory Complications in Obese Patients Planned for Laparoscopic Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University Pendik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, dilara gocmen, Dilara Göçmen, Department of Anesthesiology and Reanimation, Marmara University Pendik Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Marmara üniversitesi
Record Dates: First submitted 2025-04-16; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Obesity; Postoperative Bariatric Surgery; Laparoscopic Surgery; Individualized PEEP Treatment Strategy
Keywords: individualized PEEP treatment surgery; obesity; postoperative pulmonary complications; laparoscopic surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: this study is a double-blind study. the patient and the specialist physician performing the postoperative lung ultrasound will not know which group the patient is in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group PEEP8 (No Intervention): The first group (group PEEP8) will be applied with a fixed PEEP of 8cmH20 throughout the intraoperative period by adjusting the tidal volume of 6-8 ml/kg according to the ideal weight, and a manual recruitment maneuver (with a pressure of 30 cmH2O for 40 seconds) will be applied after the pneumoperitoneum is terminated.
- group DC (Experimental): The second group (Group DC) will be ventilated in VCV mode again and a tidal volume of 6-8 ml/kg will be given according to their ideal weight. The PEEP value at which the highest compliance value determined in the anesthesia device is obtained will be adjusted. In this group, PEEP titration will be repeated during pneumoperitoneum and skin closure. While PEEP titration is applied to the patients, a recruitment maneuver will also be applied. In this maneuver, PEEP will be increased at 2-minute intervals with a maximum peak pressure of 45 cmH2O and a driving pressure of 15 cmH2O, and when the target is reached, it will be decreased and the PEEP value will be adjusted at the value at which the highest compliance is obtained.
  Interventions: Procedure: dynamic compliance guided PEEP titration

INTERVENTIONS:
Procedure: dynamic compliance guided PEEP titration — In order to find the individualized optimal PEEP value, PEEP will be increased at 2-minute intervals with a maximum peak pressure of 45 cmH2O and a driving pressure of 15 cmH2O. Recruitment will be performed. When the target is reached, the PEEP value will be adjusted to the value at which the highest dynamic compliance is achieved by decreasing it.
  Arms: group DC

SUMMARY:
This study aims to investigate the effects of the personalized application of respiratory pressures applied to patients undergoing laparoscopic bariatric surgery when they are connected to a ventilator under general anesthesia, on the postoperative period. The effects of the ventilation practices that are fixed in routine practice and revised according to various variables during the surgery during artificial respiration after intubation under general anesthesia will be examined with ultrasonography. No change will be made to the routine anesthesia practice for this purpose, the pressure values in the ventilator under general anesthesia will be adjusted during the surgery within the framework of the values used in anesthesia practice. After the surgery, the lung area will be examined with ultrasound in the recovery unit and the findings will be recorded. This study does not have any undesirable effects or risks. This study does not include any interventional procedures.

DETAILED DESCRIPTION:
Our study is a double-blind study and the specialist physician performing the postoperative lung ultrasound will not know which group the patient is in. Before the patients are taken into surgery, they will be determined by a permanent anesthesiologist in the preoperative evaluation room using the closed envelope method. The teams that perform all measurements and randomize the patients will remain constant throughout the study. Patients who agree to participate in the study will undergo standard monitoring (heart rate - HR, peripheral oxygen saturation - SpO2, noninvasive blood pressure - NIBP, end-tidal carbon dioxide pressure - etCO2) followed by anesthesia induction. After endotracheal intubation, patients will begin to breathe with volume-controlled ventilation-VCV mode.

In the first group (group PEEP8), a tidal volume of 6-8 ml/kg will be adjusted according to their ideal weight and a fixed PEEP of 8cmH20 will be applied throughout the intraoperative period, and a manual recruitment maneuver (with a pressure of 30 cmH2O for 40 seconds) will be applied after the pneumoperitoneum is terminated. The second group (Group DC) will be ventilated in VCV mode again and a tidal volume of 6-8 ml/kg will be given according to their ideal weight. The PEEP value at which the highest compliance value determined in the anesthesia device is obtained will be adjusted. In this group, PEEP titration will be repeated during pneumoperitoneum and skin closure. While applying PEEP titration to patients, a recruitment maneuver will also be applied. In this maneuver, PEEP will be increased at 2-minute intervals so that the maximum peak pressure is 45 cmH2O and the driving pressure is 15 cmH2O, and when the target is reached, it will be decreased and the PEEP value will be adjusted at the value at which the highest compliance is obtained. The spO2 values of the patients in both groups will be targeted as 92-94%, the EtCO2 values as 35-45 cmH2O, and the FiO2 and respiratory rate will be adjusted accordingly. After extubation, the patient will be taken to the recovery room and monitored. After 15 minutes, lung ultrasound (USG) will be performed on patients in both groups by an experienced anesthesiologist who is blinded to the study using the MyLab ™ Seven convex probe (2-5 MHz). Both hemithoraxes will be divided into 6 regions by 3 vertical lines from the anterior axillary, parasternal and posterior axillary lines; 2 horizontal imaginary lines 1 cm above the nipple and at the level of the diaphragm. Each region will be evaluated for lung sliding movement, A lines, B lines, consolidation, air bronchograms, pleural effusion and pneumothorax, and the total score calculated using the modified lung ultrasound score will be recorded and compared.

ELIGIBILITY:
Inclusion Criteria:

- Patients over the age of 18, with a body mass index of 35 and above, and who are scheduled for laparoscopic bariatric surgery will be included in our study.

Exclusion Criteria:

* Patients with advanced COPD,
* Patients with a history of pneumothorax,
* Patients with lung bullae,
* Patients who have undergone thoracic surgery,
* Patients with a diagnosis of major cardiac disease (valve diseases, heart failure, systolic dysfunction),
* Patients with severe respiratory failure,
* Patients with previous pulmonary surgery will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Modified lung ultrasound score | At the end of the surgery, a modified lung ultrasonography will be performed in the recovery unit.
  Each hemithorax will be divided into 6 regions by 3 vertical lines from the anterior axillary, parasternal and posterior axillary lines; 2 horizontal imaginary lines 1 cm above the nipple and at the level of the diaphragm. Each region will be evaluated in terms of lung sliding motion, A lines, B lines, consolidation, air bronchograms, pleural effusion and pneumothorax, and the total score calculated for 12 regions will be recorded and compared using the scoring system defined by Monastesse et al (2017).

SECONDARY OUTCOMES:
postoperative pulmonary complications | postoperative 3 days
  Patients will be visited daily during the postoperative period and evaluated for oxygen need, non-invasive CPAP need, saturation values, pneumonia, shortness of breath, and respiratory distress.
hospitalization day | postoperative day 1-8
  The number of days postoperatively, the number of days spent in intensive care or in the patient room will be recorded.
postoperatif blood result | postoperative day 1 to 8
  Postoperative white blood cell, neutrophil, CRP, creatine values will be recorded.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Marmara University Pendik Training and Reseach Hospital, Istanbul, Pendik
  - Marmara University Pendik Training and Research Hospital, Istanbul, pendik

IPD SHARING:
Plan to Share IPD: No
It will be shared once enough data has been accumulated.

REFERENCES:
- See also: This study shows that LUS is highly feasible and frequently detects postoperative pulmonary complications after major abdominal surgery. — https://pubmed.ncbi.nlm.nih.gov/31523784/